CLINICAL TRIAL: NCT05848167
Title: Senile Osteoporotic Fractures Cohort Study
Brief Title: Senile Osteoporotic Fractures Cohort Study（SOFCS）
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Suzhou Municipal Hospital (Other)
Responsible Party: Principal Investigator, Mo Zhou, Director, Suzhou Municipal Hospital
Other Study IDs: GSKY20210404
Record Dates: First submitted 2023-04-26; First posted 2023-05-08 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Osteoporotic Fractures
Keywords: Senile osteoporotic fracture,Cohort study,mechanism,outcome
MeSH Terms: conditions — Osteoporotic Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Osteoporotic fracture is one of the main causes of disability and death in elderly patients. Specific disease cohort study is an important basis for accurate prevention and treatment of senile osteoporotic fractures. Investigators plan to collect and manage the baseline and clinical information of more than 2000 elderly patients with osteoporotic fractures after surgery through the platform of special disease collaborative prevention and treatment system and medical record database of Suzhou Municipal Hospital in two years, and carry out short-term and long-term follow-up observation.

DETAILED DESCRIPTION:
Osteoporotic fracture is one of the main causes of disability and death in elderly patients. Compared with patients with no history of fractures, the risk of a second fracture after an initial fracture doubled, with a fatality rate of up to 34.8%. There has been a lot of progress in the diagnosis and treatment of osteoporotic fractures in the elderly. However, there are few reports on the diagnosis and treatment of osteoporotic fractures in the elderly after surgery. Based on previous studies, it is found that the re-fracture after operation of osteoporotic fracture in the elderly is not only directly caused by the fall, but also caused by the interaction of multiple risk factors including environmental factors, physiological factors and neuroskeletal musculoskeletal system. Therefore, it is of great significance to break the traditional diagnosis and treatment mode, improve the diagnosis and treatment effect, and save medical resources to carry out research on the disease characteristics, rules and risk warning after senile osteoporotic fracture operation. Specific disease cohort study is an important basis for accurate prevention and treatment of senile osteoporotic fractures. Investigators plan to collect and manage the baseline and clinical information of more than 2000 elderly patients with osteoporotic fractures after surgery through the platform of special disease collaborative prevention and treatment system and medical record database of Suzhou Municipal Hospital in two years, and carry out short-term and long-term follow-up observation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥65 years old
2. Patients with osteoporosis
3. No gender limitation

Exclusion Criteria:

1. < 65 years old;
2. Non-osteoporotic fracture;
3. Alzheimer's disease;
4. Bone tumors.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Elderly patients after operation of osteoporotic fracture.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2024-05-14 (Estimated); Study Completion 2024-07-14 (Estimated)

PRIMARY OUTCOMES:
Bone mineral density | two years
  BMD

CONTACTS AND LOCATIONS:
Overall Officials: Hao Y feng, doctor, Study Chair — Suzhou Municipal Hospital
Locations (1):
- Suzhou Municipal Hospital, Suzhou, Jiangsu, China